CLINICAL TRIAL: NCT01788254
Title: Open Label Study for the Functional Characterization of Drug Metabolism and Transport
Acronym: IKP243
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Matthias Schwab (Other)
Responsible Party: Sponsor-Investigator, Matthias Schwab, Prof. M.D., University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IKP243; 2011-002291-16 (EudraCT Number)
Record Dates: First submitted 2013-01-31; First posted 2013-02-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Genotype-related Drug Metabolism
Keywords: pharmacokinetic/genetic; Cyp450 polymorphisms; Noninvasive functional characterization of liver heart and kidneys using MRI
MeSH Terms: interventions — Codeine; Midazolam; Pravastatin; talinolol; Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug cocktail (Experimental): A single oral low dose of codeine 5 mg and midazolam 1 mg administered as drop, pravastatin 5 mg, talinolol 2.5 mg, and torsemide 0.25 mg provided in capsules will be given together at the same time point (cocktail).
  Interventions: Drug: Codeine; Drug: Midazolam; Drug: pravastatin; Drug: Talinolol; Drug: torsemide

INTERVENTIONS:
Drug: Codeine — A single oral low dose of codeine 5 mg and midazolam 1 mg administered as drop, pravastatin 5 mg, talinolol 2.5 mg, and torsemide 0.25 mg provided in capsules will be given together at the same time point (cocktail).
Drug: Midazolam — A single oral low dose of codeine 5 mg and midazolam 1 mg administered as drop, pravastatin 5 mg, talinolol 2.5 mg, and torsemide 0.25 mg provided in capsules will be given together at the same time point (cocktail).
Drug: pravastatin — A single oral low dose of codeine 5 mg and midazolam 1 mg administered as drop, pravastatin 5 mg, talinolol 2.5 mg, and torsemide 0.25 mg provided in capsules will be given together at the same time point (cocktail).
Drug: Talinolol — A single oral low dose of codeine 5 mg and midazolam 1 mg administered as drop, pravastatin 5 mg, talinolol 2.5 mg, and torsemide 0.25 mg provided in capsules will be given together at the same time point (cocktail).
Drug: torsemide — A single oral low dose of codeine 5 mg and midazolam 1 mg administered as drop, pravastatin 5 mg, talinolol 2.5 mg, and torsemide 0.25 mg provided in capsules will be given together at the same time point (cocktail).

SUMMARY:
Aim of this study is to comprehensively assess in healthy volunteers the metabolic processes and factors that define drug response. Sources of variability are to be investigated and factors that can alter the hepatic metabolism and the pharmacokinetics of drugs shall be quantified.

Determination of variability is important when the pharmacokinetics of new drugs is being investigated and when the concept of individualized medicine is to be further developed. It is important to identify and differentiate between pharmaceutical, physiological (e.g. liver blood flow, renal function), environmental (e.g. foods and lifestyle), and genetic sources of inter-individual variability. For instance, inaccurate or false conclusions may be drawn from a single pharmacokinetic study, if the investigated medicine is metabolized by an enzyme with large inter-individual variability. Knowing the causes of variability and of the quantitative contribution of various processes might help to improve the oral formulations of drugs, might help selecting the right preclinical tests and selection criteria during clinical development, provide the basis to understand the influence of disease and to optimize established drug treatments in order to make future drug treatment safer and more efficient.

This study is designed as an add-on to the study "TWINS: Open Label Repeated Dose Study for the Evaluation of Heritability of and Genetic Influences on Drug Pharmacokinetics" (Eudra-CT: 2008-006223-31). Twins are not a random sample of the population, and they differ in their developmental environment. In this sense they are not representative for the population Thus, the results of TWINS cannot be automatically generalized but instead require validation in a representative population sample. While both studies assess pharmacologic factors important for drug response, TWINS contributes in particular data on the heritability of these processes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to study entry including informed consent for genetic research
* Both genders (male and female)
* Healthy adults aged ≥18 to <65 years
* Bodyweight not less than 48 kg and not more than 120 kg. BMI not less than 18 kg/m² and not greater than 33 kg/m².
* Smokers and nonsmokers. Smoking siblings will only be included if both siblings are smoking to a similar extend (+/- 10 cigarettes per day)
* healthy volunteers
* Dizygotic twins will only be included if both siblings are of the same gender, either male or female and triplets, quadruplets or other multiplets if at least two siblings of the same gender are considered.

Exclusion Criteria:

* Participation in a clinical trial involving the administration of medicines during the last 30 days or use of any other investigational or non-registered drug or vaccine during the study period or within 30 days preceding the first dose of study drugs
* Blood, plasma or thrombocyte donation during the last 30 days prior to application of the test drugs.
* Pregnancy or lactation period
* Any relevant clinical and pathological findings at physical examination, ECG, taking blood pressure or in clinical chemistry tests (deviation of more than 10% of the normal range).
* Positive signal from urinary drug test
* Raynaud's syndrome
* Taking any medication within 7 days before or during the trial with the following exceptions: Single doses of mild analgesics (e.g. aspirin, paracetamol, ibuprofen) an oral contraceptives.
* History of severe hypersensitivity reactions and anaphylaxis.
* History of intolerance or allergic reactions to or contraindication for any of the investigational products.
* Clinically significant diseases as judged by the investigator.
* Contraindication against MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Blood levels and clearance (dose/AUC) of midazolam | 8 hours
Blood levels and clearance (dose/AUC) of torsemide | 8h
Blood levels and clearance (dose/AUC) of codeine | 8h
Blood levels and clearance (dose/AUC) of talinolol | 8h
Blood levels and clearance (dose/AUC) of pravastatin | 8h

SECONDARY OUTCOMES:
determine metabolite profile | 8 hours
  To determine metabolite profile of the phenotyping probes and to assess Pharmacokinetic parameters and/or metabolic ratios in relation to underlying genotypes as well as to validate the heritability estimates derived from TWINS.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schwab, Prof., M.D., Principal Investigator — Dr. Margarete Fischer Bosch Institute of Clinical Pharmacology and University of Tuebingen
Locations (2):
- Germany (2):
  - Dr. Margarete Fischer-Bosch-Institute of Clinical Pharmacology, Stuttgart
  - Abteilung Klinische Pharmakologie, Tübingen